CLINICAL TRIAL: NCT03717896
Title: Thiamine As Adjunctive Therapy for Diabetic Ketoacidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Michael Donnino, Associate Professor of Medicine and Emergency Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018P000475; 1R01DK112886-01A1 (NIH)
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Diabetic Ketoacidosis
Keywords: diabetic ketoacidosis; DKA; thiamine; acidosis; oxygen consumption; lactate
MeSH Terms: conditions — Diabetic Ketoacidosis; Acidosis | interventions — Thiamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thiamine (Experimental): 200mg IV thiamine in 50mL 0.9% saline twice daily for 2 days
  Interventions: Drug: 200mg IV thiamine in 50mL 0.9% saline
- Placebo (Placebo Comparator): 100mL 0.9% saline twice daily for two days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 200mg IV thiamine in 50mL 0.9% saline — Thiamine 200mg IV every 12 hours for 2 days
  Other Names: Vitamin B1
  Arms: Thiamine
Drug: Placebo — 50mL 0.9% saline
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled trial to determine if administration of intravenous thiamine will lead to quicker resolution of acidosis in patients admitted to the hospital with diabetic ketoacidosis. The investigators will secondarily investigate whether thiamine improves cellular oxygen consumption, shortens intensive care unit (ICU) and hospital stay or decreases hospital resource utilization.

DETAILED DESCRIPTION:
Thiamine (vitamin B1) is a water-soluble vitamin that plays a key role in aerobic glucose metabolism. Thiamine is a cofactor of pyruvate dehydrogenase (PDH), an enzyme that must be activated for entry into the Krebs Cycle for aerobic metabolism. PDH activity is reduced in thiamine deficient states, resulting in a shift in pyruvate metabolism to the anaerobic pathway. This leads to increased lactate production and acidosis. Thiamine loss in the urine, with consequent thiamine deficiency, is not uncommon in diabetes. The investigators' preliminary studies have found that thiamine deficiency in occurs in as many as 39% of patients with DKA, and that thiamine levels are inversely associated with lactate and acidosis. The investigator hypothesizes that treating DKA patients with intravenous thiamine will lead to faster resolution of acidosis and improved aerobic metabolism. The investigator's secondary hypothesis is that thiamine treatment will shorten stays in the ICU and hospital and lead to utilization of fewer hospital resources.

In this randomized, double-blind, placebo-controlled trial, patients admitted to the hospital with DKA who are enrolled in the study will be randomized to either intravenous thiamine (200mg in 0.9% saline) twice daily for two days or an identical volume of 0.9% saline on the same schedule. The investigator's primary outcome is change in bicarbonate over the 24 hours following enrollment, with measurements at 0, 6, 12, 18, 24 hours, using a linear mixed-effects model. Secondarily, patients will be stratified by Type I and Type II DM. Additionally, a pre-planned sub-analysis of thiamine deficient subjects will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Bicarbonate ≤15 mEq/L
* Anion gap > 12 mEq/L
* Blood pH≤ 7.24 (if already obtained by clinical team)
* Urine ketones (qualitative) or serum ketones (β-hydroxybutyric acid) > 3 mmol/L
* Enrollment within 6 hours of presentation

Exclusion Criteria:

* Current thiamine supplementation ≥ 6 milligrams per day (i.e., more than a multivitamin)
* Competing causes of severe acidosis including seizure, carbon monoxide poisoning, cyanide toxicity, cardiac arrest, liver dysfunction (specifically defined as known cirrhosis)
* Known allergy to thiamine
* Competing indication for thiamine administration as judged by the clinical team (e.g., significant alcohol use)
* Research-protected populations (pregnant women and prisoners)
* Patient enrolled previously in same study
* Code status of Do Not Resuscitate/Do Not Intubate (DNR/DNI) or Comfort Measures Only (CMO)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
plasma bicarbonate levels | 24 hours
  Our primary outcome is change in bicarbonate over the 24 hours following enrollment with measurements at 0, 6, 12, 18, 24 hours using a linear-effects model

SECONDARY OUTCOMES:
anion gap | 24 hours
  Our secondary outcomes include change in anion gap over the 24 hours following enrollment with measurements at 0, 6, 12, 18, 24 hours using a linear-effects model
lactate | 24 hours
  Another secondary outcome is change in lactate over the 24 hours following enrollment with measurements at 0, 6, 12, 18, 24 hours using a linear-effects model
oxygen consumption by circulating mononuclear cells | 24 hours
  Oxygen consumption by circulating mononuclear cells is an index of whole body oxidative glucose metabolism. It also reflects whole body thiamine status due to the critical cofactor role of thiamine in oxidative metabolism. Mononuclear cell oxygen consumption will be assessed by the investigators when the patient is admitted into the study and again after 24 hours to determine if there is a difference between the two groups.
ICU length of stay | 24 hours
  ICU length of stay reflects how rapidly the patient recovers from the most severe consequences of diabetic ketoacidosis. The investigators will record this parameter from hospital records.to determine if there is a difference between the two groups.
hospital length of stay | 24 hours
  Hospital length of stay reflects how long it takes a diabetic ketoacidosis patient to recover to the point where he/she can be released from the hospital. The investigators will record this parameter from hospital records to determine if there is a difference between the two groups.
hospital resource usage | 24 hours
  The investigators will record this parameter from hospital records to determine if there is a difference between the two groups

OTHER OUTCOMES:
SOFA score (sequential organ failure assessement score) | 24 hours
  Investigators will assess the difference between the thiamine and placebo groups in SOFA score.
  The SOFA score will be defined using a modification in which the arterial oxygen saturation/fraction of inspired oxygen (SaO2 /FiO2) ratio is substituted for the partial pressure of arterial oxygen/fraction of inspired oxygen (PaO2 /FiO2 ratio).
C-peptide levels | 0 and 72 hours
  Investigators will measure C-peptide levels at time of study drug administration and at 72 hours or before discharge. This outcome will be analyzed separately for patients with diabetes type 1 and type 2.
Duration of insulin therapy | First 7 days after enrollment
  The duration of insulin therapy is calculated by examining the hospital clinical information systems for all records of IV insulin infusion beginning at the time of enrollment. The start and the stop time-stamps of medication infusion are used to calculate a duration of infusion.
Cognitive function: Hopkins Verbal Learning Test | between 72 and 96 hours after enrollment or prior to discharge (whichever comes first)
  As an exploratory outcome, we will measure cognitive function using the Hopkins Verbal Learning Test (measures verbal learning and memory). The test will be administered by trained research assistants at the patient's bedside 72-96 hours after enrollment or prior to discharge (whichever comes first).
Cognitive function: Brief Visual Spatial Memory Test | between 72 and 96 hours after enrollment or prior to discharge (whichever comes first)
  As an exploratory outcome, we will measure cognitive function using the Brief Visual Spatial Memory Test (measures visuospatial memory). The test will be administered by trained research assistants at the patient's bedside 72-96 hours after enrollment or prior to discharge (whichever comes first).
Cognitive function: Trail Making Test A and B | between 72 and 96 hours after enrollment or prior to discharge (whichever comes first)
  As an exploratory outcome, we will measure cognitive function using the Trail Making Test A and B (measurement of cognitive function utilizing connection of dots by correct order). The test will be administered by trained research assistants at the patient's bedside 72-96 hours after enrollment or prior to discharge (whichever comes first).
Cognitive function: WAIS-IV Digit Span | between 72 and 96 hours after enrollment or prior to discharge (whichever comes first)
  As an exploratory outcome, we will measure cognitive function using the WAIS-IV Digit Span (measures working memory). The test will be administered by trained research assistants at the patient's bedside 72-96 hours after enrollment or prior to discharge (whichever comes first).
Cognitive function: Test of Verbal Fluency and Animal Naming | between 72 and 96 hours after enrollment or prior to discharge (whichever comes first)
  As an exploratory outcome, we will measure cognitive function using the Test of Verbal Fluency and Animal Naming (measures phonemic and semantic verbal fluency). The test will be administered by trained research assistants at the patient's bedside 72-96 hours after enrollment or prior to discharge (whichever comes first).
Cognitive function: Test of Premorbid Functioning | between 72 and 96 hours after enrollment or prior to discharge (whichever comes first)
  As an exploratory outcome, we will measure cognitive function using the Test of Premorbid Functioning (estimates premorbid intellectual function). The test will be administered by trained research assistants at the patient's bedside 72-96 hours after enrollment or prior to discharge (whichever comes first).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Donnino, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vine J, Mehta S, Balaji L, Berg KM, Berlin N, Liu X, Ngo L, Shea M, Moskowitz A, Donnino MW, Grossestreuer AV. Thiamine as adjunctive therapy for diabetic ketoacidosis (DKAT) trial protocol and statistical analysis plan: a prospective, single-centre, double-blind, randomised, placebo-controlled clinical trial in the USA. BMJ Open. 2024 Feb 29;14(2):e077586. doi: 10.1136/bmjopen-2023-077586. PMID 38423765